CLINICAL TRIAL: NCT00715715
Title: A Pilot Study of Adefovir Dipivoxil Alone and After Prednisone Priming for the Treatment of Asian Patients With HBeAg-positive Chronic Hepatitis B
Brief Title: Efficacy Study of Prednisone Priming to Treat Asian Chronic Hepatitis B Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn studies.
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Principal Investigator, Ting-Hui Hsieh, Attending, Gastroenterology, Maimonides Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-01-IVA6
Record Dates: First submitted 2008-07-11; First posted 2008-07-15 (Estimated); Last update posted 2012-04-20 (Estimated); Status verified 2012-04

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B e Antigen; HBeAg-positive chronic hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): Patients that meet the requirements listed above will be selected sequentially. Blood tests, including liver function tests and hepatitis profiles will be taken. A liver biopsy will be done before the treatment to evaluate the severity of hepatitis.
  For randomly selected patients not treated with steroids: The patients will receive 6 weeks of sugar pills (placebo) before taking Adefovir dipivoxil (Hepsera) 10 mg daily for a minimum of 52 weeks.
  All patients will get another liver biopsy at week 48 to evaluate the improvement of liver inflammation after their treatment. Blood tests will be drawn in accordance with the standard treatment. Generally speaking, hospitalization is not required for this study.
- 2 (Experimental): Patients that meet the requirements listed above will be selected sequentially. Blood tests, including liver function tests and hepatitis profiles will be taken. A liver biopsy will be done before the treatment to evaluate the severity of hepatitis.
  For randomly selected patients treated with steroids: The patients will receive prednisone 30 mg daily for 3 weeks, 15 mg daily for 1 week, no treatment for 2 weeks, followed by Adefovir dipivoxil (Hepsera) 10 mg daily for a minimum of 52 weeks.
  All patients will get another liver biopsy at week 48 to evaluate the improvement of liver inflammation after their treatment. Blood tests will be drawn in accordance with the standard treatment. Generally speaking, hospitalization is not required for this study.
  Interventions: Drug: Prednisone Priming

INTERVENTIONS:
Drug: Prednisone Priming — For randomly selected patients treated with steroids: The patients will receive prednisone 30 mg daily for 3 weeks, 15 mg daily for 1 week, no treatment for 2 weeks, followed by Adefovir dipivoxil (Hepsera) 10 mg daily for a minimum of 52 weeks.
  Arms: 2

SUMMARY:
Patients with chronic hepatitis B constantly produce the virus in the body. The disease of chronic hepatitis B is the body responding to the virus. Use of steroids can adjust this response. After taking steroids, viral production usually increases and liver function tests increase. After stopping steroids, viral production usually decreases. Many studies in the past have studied taking a low dose steroid before treating hepatitis B. Those studies have shown that low dose steroids help your body to clear the virus. The goal of this study is to improve the liver function by slowing viral growth.

DETAILED DESCRIPTION:
Asian patients who are older than 16 years of age and have HBeAg-positive chronic hepatitis B and good liver function will be entered in this study. Qualified patients also have positive hepatitis B surface antigen (HBsAg) for at least 24 weeks before screening, evidence of chronic hepatitis on a baseline liver-biopsy sample obtained within 52 weeks before entry, evidence of HBV DNA by any commercial tests at least 4 weeks before screening, an high HBV DNA level (at least 20,000 IU/mL) at screening, and a high serum ALT level (1.0 to 5.0 times the upper limit of normal) at screening.

This study involves experimental use of an approved drug (Prednisolone) on chronic hepatitis B patients. Patients will be involved in the study for up to 96 weeks from enrollment. There is no external sponsor, commercial sponsor nor federal agency on this study. The study will be conducted only at Maimonides Medical Center, its GI clinic and faculty practice. About 40 subjects will be involved in the study overall. All the subjects will be filled up locally.

ELIGIBILITY:
Inclusion Criteria:

This study is seeking patients with the following:

* Asians older than 16 years of age
* HBeAg-positive chronic hepatitis B, and
* Good liver function
* Positive hepatitis B surface antigen (HBsAg) for at least 24 weeks before screening
* Liver biopsy in the past year showing of chronic hepatitis
* Blood testing showing HBV DNA in the past 4 weeks before screening
* Blood test showing high HBV DNA level (at least 20,000 IU/mL); AND
* Liver function test showing high serum ALT level (1.0 to 5.0 times the upper limit of normal).

Exclusion Criteria:

* Ongoing drug abuse
* Active alcoholism
* Coinfection with hepatitis C, hepatitis D, or HIV
* Presence of other forms of liver disease
* Use of interferon alfa, thymosin, or antiviral agents with activity against hepatitis B within 24 weeks before randomization
* Prior lamivudine therapy lasting more than 12 weeks
* Previous treatment with Adefovir dipivoxil
* AFP level greater than 100 ng/mL
* Decompensated liver disease
* History of ascites requiring diuretics or paracentesis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The primary efficacy end points at week 48 include the reduction in HBV DNA, HBeAg seroconversion, normalization of ALT. | week 48

SECONDARY OUTCOMES:
Secondary efficacy end point is the proportion of patients with histologic improvement. | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Li, MD, Principal Investigator — Maimonides Medical Center; Ting-Hui Hsieh, MD, Principal Investigator — Maimonides Medical Center
Locations (1):
- Maimonides Medical Center, Brooklyn, New York, United States